CLINICAL TRIAL: NCT02859610
Title: Characterization of Microparticles in Cirrhosis and Portal Hypertension With Implications
Brief Title: Microparticles in Cirrhosis and Portal Hypertension
Acronym: MicroCir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-A01258-37
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Liver Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cirrhotic patients (Other): We prospectively included 90 cirrhotic patients .
  Interventions: Other: research on interactions between portal hypertension and microparticles
- healthy volunteers (Other): The pilot cohort was compared with 10 healthy volunteers.
  Interventions: Other: research on interactions between portal hypertension and microparticles

INTERVENTIONS:
Other: research on interactions between portal hypertension and microparticles

SUMMARY:
research on interactions between portal hypertension and microparticles

DETAILED DESCRIPTION:
It has already been shown that increased certain markers of stress, such as prolonged elevation of CRP in the absence of bacterial infection, increased free cortisol and serum copeptin, are associated with an excess of mortality in cirrhosis.

MPs are membrane vesicles of variable size between 0.1 and 1 .mu.m, released into the extracellular space following activation or cellular apoptosis. MPs are also found in the circulating blood of healthy volunteers and their plasma levels rise in certain diseases to increased thrombotic risk, such as in cancer. Their membrane is composed of antigens whose organization is characteristic of the parent cell and negatively charged phospholipids, phosphatidylserines, conferring pro-coagulant properties to these MPs.

Currently, work on the MPs are increasing following the discovery of their involvement in physiological processes such as proliferation, differentiation, cell activation and immune response but it is certainly their pro-thrombogenic power that was the most studied.

Recent studies have also implicated MPs in the pathophysiology of chronic liver disease. Cirrhotic patients have elevated concentrations of MPs from leukocytes, endothelial cells and hepatocytes compared to control subjects, and concentrations of MPs increase with worsening liver function. Increasing MPs during the cirrhosis may be related on the one hand with a decreased clearance and secondly with an excess of proinflammatory cytokines by increasing the phenomenon of intestinal bacterial translocation. The assumption of the role of systemic inflammation in the training of MPs is reinforced by the existence of a significant correlation between the original MPs hepatocyte or buffy endothelial and CRP Thus, the increase in MPs observed with the increase of PH could increase the risk of thrombosis in intestinal microcirculation leading to enterocytic suffering from ischemic, reflected by an increase in serum concentrations of I-FABP ( intestinal fatty acid binding protein). This suffering enterocytes leads to increased intestinal bacterial translocation and ultimately to increased formation of MPs. These MPs could also worsen liver function by the same phenomenon of thrombosis in the hepatic microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* Non infected cirrhotic patient (30 patients Child-Pugh A, 30 Child-Pugh B et 30 Child-Pugh C).
* 10 heathly volunteer (groupe contrôle).

Exclusion Criteria:

* legal incapacity or limited legal capacity
* Subject unlikely to cooperate in the study and / or low early cooperation by the investigator
* Subject without health insurance
* Pregnant woman
* About being in the disqualification of another study or under the "national register of volunteers."
* Any proven or suspected infection
* Pre-hepatic portal hypertension (door thrombosis) or post-liver (Budd-Chiari) transplant patients, HIV infection (also refusing HIV status) or patients on immunosuppressive therapies (including corticosteroids) interferon taken
* Treatment with anticoagulants or antiplatelet upper gastrointestinal bleeding in the two months prior
* Patients with TIPS
* Any cancer pathology proven and current.
* Chronic heart failure (stage III or IV of the classification of the New York Heart Association [NYHA])
* Inability to receive clear information in patients with severe encephalopathy and do not have someone you trust

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Level of expression of microparticles in cirrhotic patients with hepatic function of varying severity (Child- Pugh A to C) and in 10 healthy controls. | one year
Procoagulant activity of microparticles in cirrhotic patients with hepatic function of varying severity (Child- Pugh A to C) and in 10 healthy controls. | one year